CLINICAL TRIAL: NCT05146375
Title: Genes Modulating the Severity of Aortic Aneurysms (MSF1-TGFBR2)
Acronym: MSF1-TGFBR2
Status: Active, not recruiting | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Fédération Française de Cardiologie (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-02
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Vascular Diseases, Aneurysm; TGFBR2 mutation
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Vascular Diseases; Aneurysm | interventions — Receptor, Transforming Growth Factor-beta Type II

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample (serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MSF1: Each member of the MSF1 family who consents to participate to the study will be included.
  Interventions: Biological: TGFBR2

INTERVENTIONS:
Biological: TGFBR2 — TGFBR2 mutation correlation with severity of the aortic disease. Blood sampling. Serum will be analysed by DNA sequencing to detect specific mutations involved in aneurysms.
  Cutaneous biopsy. Fibroblast culture will be done to assess the transcriptome analysis.

SUMMARY:
This project concerns a population at risk of sudden death by dissection of the thoracic aorta. Its interest is to make it possible to recognize the genes that protect or worsen the evolution of aneurysms, to better understand the mechanisms involved, to detect and treat aneurysms of the thoracic aorta, wich is a pathology that is completely silent clinically until life-threatening complications.

The variability in the severity of the disease within the same family is related to modifier genes.

The objective is to find the modifying factors that account for the variability in the severity of the progression of aneurysms of the thoracic aorta.

DETAILED DESCRIPTION:
Thoracic aortic aneurysms are silent, asymptomatic, potentially fatal pathologies due to the risk of aortic dissection. More and more often they are found during imaging tests done for another reason. Some aneurysms have genetic origin (autosomal dominantly inherited) and are particularly interesting because they can be recognized early (due to possible family screening), which allows us to understand the natural history of this pathology. The discovery of genes whose mutations explain the occurrence of these family aneurysms (initiator gene) has also made it possible to improve family screening and to better understand the pathophysiology of these aneurysms: we now recognize 3 groups of genes involved (extracellular matrix, contractile proteins of smooth muscle cell, TGF-β pathway (Transforming Growth Factor) [including mutations in TGF-β receptor 2 gene, TGFBR2]).

The variability in the severity of signs and aortic involvement is particularly marked in patients with aortic aneurysms due to mutations in the TGFBR2 gene. Some patients with these mutations present aggressive aneurysms with early dissection. Other patients have isolated late-onset aneurysms, and others have no signs.

This variability generates problems for clinical practice to give appropriate genetic advice, but also to adapt imaging monitoring, therapy, or sports restriction.

The present protocol aims is to investigate the variability in the severity of the disease within a large family carrying a mutation in the TGFBR2 gene. The MFS1 family is a family in which the aortic pathology is due to a mutation in the TGFBR2 gene. All patients with this family carry the same TGFBR2 mutation, heterozygous.

ELIGIBILITY:
Inclusion Criteria:

Member of MSF1 family. The MFS1 family is a family in which the aortic pathology is due to a mutation in the TGFBR2 gene. All patients with this family carry the same TGFBR2 mutation (heterozygous)

Exclusion Criteria:

Refusal or linguistic or psychological inability to sign informed consent

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 53 members of the MFS1 family are currently identified and have a medical follow-up in the national referral center for Marfan syndrome of the hospital Bichat-Claude Bernard, Paris.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical phenotype | day 1
  The criterion of severity of aortic disorder is based on the maximal aortic diameter measurement (in millimeter, measured at the level of the sinuses of Valsalva) and on age-adjusted aortic dilation.

SECONDARY OUTCOMES:
TGFBR2 and other gene mutations involved in aneurysms | All samples will be analysed at the same time, at the end of the recruitment.
  correlation genotype/phenotype
Genotype analysis | All samples will be analysed at the same time, at the end of the recruitment.
  Comparison between worst phenotype and genotype / Comparison between best phenotype and genotype
Transcriptome analysis | All samples will be analysed at the same time, at the end of the recruitment.
  Gene expression will be assessed by RNA-sequencing. Correlation between transcriptional profiles and clinical phenotype will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, MD, Principal Investigator — Hopital Bichat-Claude Bernard
Locations (1):
- Hopital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No